CLINICAL TRIAL: NCT05635513
Title: Owlet Smart Sock 3 Accuracy on Infants
Status: Completed | Type: Observational
Sponsor: Owlet Baby Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OWL NICU 07-2021
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-12

CONDITIONS: Hypoxia Neonatal
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Owlet OSS V3 — A wearable pulse oximeter designed for monitoring infants and children in a home environment

SUMMARY:
The purpose of this research study is to evaluate the Owlet Smart Sock 3 wireless pulse oximeter performance in assessing the heart rate and oxygen saturation in neonatal population, while measuring the same parameter with a standard wired pulse oximeter simultaneously. The monitoring duration with the study device will be a maximum of 60 minutes, after which the recorded data from the Owlet Smart Sock 3 and the standard wired pulse oximeters will be de-identified and analyzed.

DETAILED DESCRIPTION:
This prospective observational study compared the HR and SpO2 measurements of the OSS3 (Owlet, Utah, USA) with the Masimo SET® (Masimo Corporation, California, USA) in infants admitted to the University of Utah NICU. The inclusion criteria were infants who weighed 1.7-2.5 kg at the time of monitoring and were medically stable to tolerate routine care. The exclusion criteria were: infants with significant anomalies, congenital deformities, or medical instability. Infants with an intravenous catheter (IV) and skin lesions on either foot were excluded from the study. The wireless device being tested was the OSS3. The gold standard for validating the pulse oximeter's accuracy is arterial blood oxygen saturation (SaO 2 ) at the pulse oximeter sensor site. [6] However, obtaining SaO2 is an invasive arterial blood test for infants. To avoid this conflict, the OSS3 was tested against the reference FDA-approved wired pulse oximeter Masimo.

The study was approved by the University of Utah Institutional Review Board, and informed consent was obtained from parents. During the measurement, OSS3 and Masimo were placed on the infants with one device on each foot. Since the data obtained from the study devices can not be recorded in the hospital electronic medical record, the hospital wired pulse oximeter (Philips, Amsterdam, Netherlands) continued to be used on one of the infant's hands during the study period. OSS3 and Masimo were calibrated appropriately against the hospital wired pulse oximeter with matching HR and SpO 2 readings. Pulse oximetry data were collected simultaneously for 60 minutes on the quiet infants. The two devices (OSS3 and Masimo) continuously recorded HR (beats per minute, bpm) and SpO2 (%) every two seconds. Data from the 2 devices were uploaded and compared according to their time stamped measurements. The paired data agreement was compared using Pearson's correlation coefficient (r), Bland-Altman, Average Root Mean Square (ARMS), and Prevalence and Bias Adjusted Kappa (PABAK) analyses.

ELIGIBILITY:
Inclusion Criteria:

* Infant who weigh between 1.7kg and 2.3kg
* Infant who is admitted to U of U NICU

Exclusion Criteria:

* Infant who has injuries, deformities, abnormalities, or intravenous catheter in the extremities that may prevent proper application of device
* Infant who has unstable vital signs or clinical condition
* No parental consent
* Inability to achieve adequate fit with the OSS3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants admitted to the University of Utah NICU that weigh between 1.7kg and 2.3kg and do not meet exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Owlet Oxygen Saturation Accuracy Performance | During the monitoring period (approx. 1 hour)
  Conduct a single-arm observational study to monitor oxygen saturation (SpO2) while a standard wired pulse oximeter (WPOx) will simultaneously evaluate the same parameters in the University of Utah (U of U) Neonatal Intensive Care Unit (NICU).
Owlet Pulse Rate Accuracy Performance | During the monitoring period (approx. 1 hour)
  Conduct a single-arm observational study to monitor heart rate (HR), while a standard wired pulse oximeter (WPOx) will simultaneously evaluate the same parameters in the University of Utah (U of U) Neonatal Intensive Care Unit (NICU).

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Chan, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah NICU, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided